CLINICAL TRIAL: NCT06231589
Title: Next Generation Sequencing of Embryos for Testing the Efficacy of Advanced Sperm Selection Techniques in Males With High Teratozoospermia Index
Brief Title: PGT-A Evaluates Advanced Sperm Selection in Embryos From High Teratozoospermia Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ganin Fertility Center (Other)
Responsible Party: Principal Investigator, Mohamed Nasreldin Abdelmagied Ali, Clinical Embryologist, Ganin Fertility Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GFC-008
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Teratozoospermia; Sperm DNA Fragmentation; Infertility
Keywords: Sperm selection; Teratozoospermia index; Sperm DNA fragmentation; PGT-A; Euploidy rate
MeSH Terms: conditions — Teratozoospermia; Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): 111 Males have normal Teratozoospermia index (TZI) less than 1.6. Semen processing is done by double layer density gradient method only.
- Sperm selection group PICSI or MACS (SS-Group) (Experimental): 90 Males with high TZI and sperm selection techniques such as PICSI or MACS are performed. Semen processing is done by double layer density gradient method followed by:
  (1) In case of PICSI: adding Sperm to the dot of hyaluronan on the PICSI dish, within minutes the bound sperm are attached by their acrosome to the surface of the dot. Individual bound sperm selection is done followed by ICSI.
  or (2) In case of MACS: Semen processing is done by double layer density gradient method. The resulted pellet is labeled with annexin V microbeads followed by separation on MACS Column, the eluted fraction contains non apoptotic sperm suitable for ICSI.
  Interventions: Device: Sperm Selection
- No sperm selection group (NO SS-Group) (No Intervention): 63 Males with high TZI more than 1.8 and no sperm selection techniques are performed. Semen processing is done by double layer density gradient method only.

INTERVENTIONS:
Device: Sperm Selection — Sperm selection using physiological intracytoplasmic sperm injection (PICSI dish) or magnetic-activated cell sorting (MACS) for selecting sperm with high-quality, better morphology and lower DNA fragmentation.
  Arms: Sperm selection group PICSI or MACS (SS-Group)

SUMMARY:
In this study of 264 couples, sperm selection techniques in males with high teratozoospermia index and sperm DNA fragmentation significantly increased fertilization, blastocyst development rates, and maintained comparable embryo euploidy rates through preimplantation genetic testing, suggesting the efficiency of these techniques in improving assisted reproductive outcomes.

DETAILED DESCRIPTION:
Couples seeking infertility treatment are becoming more frequent. Paternal factor shows one of the infertility causes which may have a negative impact on reproductive outcomes. Intracytoplasmic sperm injection (ICSI) is thought to be the most effective way to treat infertility. Sperm morphology evaluation is a reliable predictor of male fertility while teratozoospermia index (TZI) is a unique expression of sperm morphological assessment. A higher rate of abnormal sperm morphology tends to have higher sperm chromosomal abnormality rates. The choice of high-quality sperm through sperm selection techniques is expected to improve ICSI outcomes. In this study, a total number of 264 couples were included and divided into 3 groups: (1) Males have normal TZI (Control group: 111 males have TZI <1.6), (2) Males with high TZI and no sperm selection techniques are performed (NO-SS group: 63 males have TZI >1.8), and (3) Males with high TZI and sperm selection techniques are performed (SS-group: 90 males have TZI >1.8). The TZI was significantly (P<0.000) higher in the NO-SS and SS-group as compared to the control group. The percentage of sperm DNA fragmentation SDF in the males of the SS group was significantly higher than the controls and NO-SS group (P=0.000). The fertilization (P=0. 039) and blastocyst development rates (P= 0. 041) are significantly higher in the SS group as compared to the NO-SS group in females aged <35. A total of 1072 embryos were tested for preimplantation genetic testing for aneuploidy using NGS, although higher SDF in the males of the SS group, the embryo euploidy rates show that there is no significant difference between the SS group (56.35±3.46%) as compared to the control group (54.54±3.24%) and the NO-SS group (57.45±4.57%). In general, we found that sperm selection techniques are efficient techniques in increasing fertilization, blastocyst development rates, and euploidy rate in males with high teratozoospermia index and sperm DNA fragmentation combined.

ELIGIBILITY:
Inclusion Criteria:

1. Males diagnosed with normal and high teratozoospermia index.
2. Males with Mild to moderate OTA (oligoteratoasthenozoospermia).
3. Males aged 18-60 years.
4. Female aged 18-40 years.
5. Case must have PGT-A for all of her blastocysts.
6. Normo responder (> 5 mature oocytes).
7. Male will have to refrain from ejaculation no less than 1 day but no greater than 3 days prior semen specimen production on day of ICSI.

Exclusion Criteria:

1. Leukocytospermia.
2. Presence of varicocele.
3. Known genetic abnormality.
4. Use of sperm or oocyte donors.
5. Use of gestational carrier.
6. Presence of any of the endometrial factors that affect embryo implantation such as hydrosalpings, adenomyosis or previous uterine infection.
7. Any contradictions to undergoing in vitro fertilization or gonadotropin stimulation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 264 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Fertilization rate | 1 day
  Defined as the proportion of fertilizaed oocytes
Blastocyst development rate | 5-6 days
  Defined as the proportion of blastocysts formed on day 5 or 6
Euploidy rate | 15 days post ICSI
  Defined as the proportion of euploid blastocysts
Aneuploidy rate | 15 days post ICSI
  Defined as the proportion of aneuploid blastocysts

SECONDARY OUTCOMES:
Blastocyst quality rate | 5-6 days
  Defined as the assessment of blastocyst quality according to Gardner's criteria into: good, fair or poor
Low mosaic rate | 15 days post ICSI
  Defined as the proportion of low mosaic blastocysts
High mosaic rate | 15 days post ICSI
  Defined as the proportion of high mosaic blastocysts

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Nasreldin, MSc., Study Chair — Ganin Fertility Center; Hanan Ramadan, PhD, Principal Investigator — Cairo University; Maiada Moustafa, PhD, Principal Investigator — Helwan University; Mohamed Abas, MBB, Principal Investigator — Cairo University; Hosam Zaki, MSc, FRCOG, Study Director — Ganin Fertility Center
Locations (1):
- Ganin Fertility Center, Cairo, Maadi, Egypt

IPD SHARING:
Plan to Share IPD: Undecided